CLINICAL TRIAL: NCT06188728
Title: Effectiveness of Lifestyle Modification in Combination With Psyllium Husk Fiber Intervention on the Metabolic Health of Centrally Obese School Teachers
Brief Title: Husk Fiber Intervention on Metabolic Health of Centrally Obese School Teachers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Peshawar (Other)
Collaborators: University of Agriculture, Peshawar (Other)
Responsible Party: Principal Investigator, Amjad Ali Bacha, Dr., University of Peshawar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UPeshawar
Record Dates: First submitted 2022-03-14; First posted 2024-01-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Metabolic Disease
Keywords: insulin resistance,; High sensitive C reactive protein; Lipid Profile; Sleep quality analysis; Abdomens and epigastric health
MeSH Terms: conditions — Metabolic Diseases; Insulin Resistance | interventions — Meals; Diet; Exercise

STUDY DESIGN:
Intervention Model Description: comparing the intervention group with the control (intervention include either lifestyle modification, psyllium husk fiber or combined intervention of lifestyle modification and psyllium husk fiber.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Control group (Placebo Comparator): Group-I comprised of 30 subjects, 15 male and 15 female. The group was assigned no intervention and kept as the control group.
  Interventions: Other: Control
- LSM group (Experimental): Group II comprised 30 subjects with the equal bifurcation of male and female. Group II was assigned the intervention of lifestyle modification (the combination of diet, physical activity, and behavior therapy)
  Interventions: Behavioral: Effect of life style modification (Diet, Behavior and physical activity)
- PSH group (Experimental): Group III comprised of 30 subjects, 15 male and 15 female. Group III was assigned the 5gm psyllium husk fiber (in swelled form) two times a day, i.e., 30 minutes before breakfast and 30 minutes before dinner.
  All the subjects in the physical demonstration were briefed about the preparation and usage of psyllium husk fiber.
  Interventions: Dietary Supplement: effect of 10 gm psyllium husk fiber twice a day, 30 minutes before breakfast and dinner
- LSM&PSH (Experimental): Group IV comprised of 30 subjects, 15 male and 15 female. Group IV was assigned both the intervention of psyllium husk fiber @ 5gm two times a day, 30 minutes before breakfast and dinner in swelled gel form with the combination of lifestyle modification
  Interventions: Combination Product: Combined effect of 10 gm Psyllium husk fiber and lifestyle modification

INTERVENTIONS:
Dietary Supplement: effect of 10 gm psyllium husk fiber twice a day, 30 minutes before breakfast and dinner — comparing the effect of psyllium husk fiber and lifestyle modification alone with the combined effect of psyllium husk fiber on metabolic health of centrally obese school teachers
  Arms: PSH group
Behavioral: Effect of life style modification (Diet, Behavior and physical activity) — To assess the effect of life style modification (Diet, Behavior and physical activity) on centrally obese school teachers
  Arms: LSM group
Combination Product: Combined effect of 10 gm Psyllium husk fiber and lifestyle modification — To evaluate the combined effect of 10 gm psyllium husk fiber in gel form, 30 minutes before breakfast and dinner along with dietary, behavioral and physical activity modification on centrally obese school teachers
  Arms: LSM&PSH
Other: Control — No intervention
  Arms: Control group

SUMMARY:
A group of 120 school teachers (male=60, female=60) was divided into four subgroups for sixteen weeks of an interventional study. One group was kept in control while the other three groups were assigned intervention. One group was assigned intervention of lifestyle modification (LSM), the other group assigned the intervention of 5 gm psyllium husk fiber (PSH) two times a day, and the third group assigned the combined intervention of LSM & PSH. Each group comprised of 30 subjects with equal gender bifurcation (15 male and 15 female).

DETAILED DESCRIPTION:
The school teachers who qualified for the initial screening and eligibility criteria were formally enrolled in the intervention. An informed consent form was signed by each subject explaining the data privacy and the subject's obligation. School teachers with lifestyle modification were advised to adhere to three major components, i.e., diet modification, physical activity, and behavioral therapy. subjects in the psyllium husk fiber group were assigned the consumption of 5gm psyllium husk fiber (in swelled form) two times a day, i.e., 30 minutes before breakfast and 30 minutes before dinner. subjects in the combined group of psyllium husk fiber and physical activity were assigned both the intervention of psyllium husk fiber @ 5gm two times a day, 30 minutes before breakfast and dinner in swelled gel form with the combination of lifestyle modification, while one group remained as control (without any intervention).

ELIGIBILITY:
Inclusion Criteria:

* School teachers aged 40-60 years (male and female)
* central obesity (where central obesity for Asians is defined as the waist circumference for men ≥ 90 cm and for women ≥ 80 cm
* with no history of any chronic disease like hypertension, Diabetes, Cardiovascular diseases, taking of any regular medication, food allergies, smoking
* physical disabilities impairing the food intake and mobility, qualified the inclusion criteria.

Exclusion Criteria:

* Pregnant or lactating female school teachers were also excluded during screening.
* Subjects with an allergy to psyllium husk fiber, history of drug abuse, or any psychological or emotional disorder that might prevent the completion of the study were also excluded.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — an equal number of males and females were enrolled in the study with similar cultural, geographical and profession background
Enrollment: 90 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Anthropometry | 16 weeks
  weight (Kg),
Lipid Profile | 16 weeks
  Triglyceride, LDL, HDL and cholesterol. unit used was mg/dl.
Sleep quality analysis | 16 weeks
  wil use Pittesburge Sleep Quality Index score (ranging from 0 to 6. where 0 reflect best sleep quality and 7 represent the worst sleep quality)
abdomen and epigastric health | 16 weeks
  Likert scale (0-7). 0 represents good health and 7 represent worst epigastric and abdominal health
height (cm) | 16 weeks
  Measure height in cm (centimeter)
Waist circumference | 16 weeks
  Measure waist circumference in cm (centimeter)
BMI | 16 weeks
  weight and height will be combine to calculate the BMI (kg/m^2)

SECONDARY OUTCOMES:
Insulin resistance | 16 weeks
  will measure insulin resistance(Molar unit)
high sensitive C reactive protein | 16 weeks
  assess the inflammation biomarkers(mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: Zia Din, PhD, Study Director — Chairman department of human Nutrition
Locations (1):
- The University of Agriculture, Peshawar, Khyberpakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
once the paper is approved and research data updated to HEC digital library
Supporting Information: CSR
Time Frame: once the research paper published
Access Criteria: through google scholar